CLINICAL TRIAL: NCT03636932
Title: RENACTIF: Reduction of the Thrombotic Phenotype in Renal Insufficiency With N-AcetylCysteine A Randomized, Double-blind, Placebo-controlled, Cross-over Trial
Brief Title: RENACTIF: Reduction of the Thrombotic Phenotype in Renal Insufficiency With N-AcetylCysteine
Acronym: RENACTIF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-71; 2018-003232-80 (EudraCT Number)
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Acetylcysteine; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (NAC) group (Active Comparator)
  Interventions: Drug: N-acetylcysteine (NAC); Biological: Blood sample
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo; Biological: Blood sample

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) — Intravenous injection of 2 gram of N-acetylcysteine (NAC) during 4 weeks, 3 times per week during the first three hours of dialysis.
  Arms: N-acetylcysteine (NAC) group
Drug: Placebo — Intravenous injection of 2 gram of Placebo during 4 weeks, 3 times per week during the first three hours of dialysis.
  Arms: Placebo group
Biological: Blood sample — Circulating tissue factor assay
Biological: Blood sample — The test of pro-coagulant activity of the tissue factor

SUMMARY:
Chronic Kidney Disease (CKD) is a known risk factor of cardiovascular morbidity and mortality.

In CKD, decline of renal function results in the accumulation of uremic toxins in blood and tissue, such as Indoxyl Sulfate (IS). IS plasma level is predictive of mortality and cardiovascular disease (CVD). Patients with CKD have increased oxidative stress and circulating tissue factor (TF) levels. In vitro, IS induces an inflammatory, pro-oxidative and pro-coagulant phenotype on endothelial cells and activates TF. N-acetylcysteine (NAC) protects endothelial cells from the effects of IS. NAC reduces oxidative stress and production of activated TF. A prospective study evaluating an oral NAC treatment versus placebo in chronic hemodialysis patients showed a better cardiovascular outcome but the physiopathology was unclear.

The hypothesis is that NAC reduces cardiovascular risk by its effect on uremic toxin-induced pro-coagulant TF production.

The primary objective is to compare the effect of NAC intravenously administered at each dialysis session (2gram on 3 dialysis sessions per week) to placebo on circulating TF levels in patients with CKD on chronic hemodialysis after 4 weeks of treatment. The objective is to show a 33% decrease in circulating tissue factor (TF) levels in the NAC group compared to the control group.

It is a randomized, double-blind, placebo-controlled crossover trial that includes chronic hemodialysis patients from La Conception Hospital (AP-HM) in Marseilles, France. This is an interventional biomedical research project.

20 patients will be included in each group and will receive during 4 weeks intravenous injection.

This study will give a pathophysiological rationale for the use of NAC to reduce thrombotic and cardiovascular risk in patients with CKD. This step will provide the rationale for a clinical trial to reduce the occurrence of major cardiovascular events with IV NAC in hemodialysis (HD) patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients regardless of the etiology of their renal insufficiency for more than 3 months on a cycle of 3 sessions per week
* Hemodialysis patients at least 4 hours per dialysis session
* Patients with a weight of more than 40 kilogram
* Patients capable of giving informed consent, agreeing to participate in the study and having signed a consent
* Patient able to understand a written questionnaire

Exclusion Criteria:

* Pregnant or lactating women
* Persons deprived of their liberty or hospitalized without consent
* Majors under legal protection or unable to express their consent
* Possibility of recovery of renal function (scleroderma for example)
* Chronic progressive infection that may affect their thrombotic risk
* Patients under 40 kilogram
* Patient taking oral anticoagulants
* Patient with a known allergy to the active molecule or to any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
compare the effect of N-acetylcysteine (NAC) intravenously administered | 12 months
  show a 33% decrease in circulating tissue factor levels in the N-acetylcysteine (NAC) group

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No